CLINICAL TRIAL: NCT04641676
Title: A Study to Examine the Value of Broad Agnostic NGS Panel Testing Versus Reimbursed Organ-directed NGS: a Belgian Precision Study of the BSMO in Collaboration With the Cancer Center
Brief Title: A Study to Examine the Value of Broad Agnostic Next Generation Sequencing (NGS) Panel Testing Versus Reimbursed Organ-directed NGS: a Belgian Precision Study of the BSMO in Collaboration With the Cancer Center
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Belgian Society of Medical Oncology (Other)
Collaborators: Foundation Medicine (Industry); Sciensano (Other Government); Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: BSMO2020-1
Record Dates: First submitted 2020-10-28; First posted 2020-11-24 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Metastatic Cancer; Local Tumor Invasion
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Foundation medicine NGS in parallel with local NGS (Other): The patient will have in parallel FMI NGS test and Local reimbursed NGS test.
  Interventions: Diagnostic Test: NGS testing
- Foundation Medicine NGS (Other): The patient will have only FMI NGS test.
  Interventions: Diagnostic Test: NGS testing
- LB Foundation Medicine NGS test (Experimental): The patient do not have enough biopsy material or have tumor not accessible for a biopsy will have a liquid biopsy Foundation Medicine test.
  Interventions: Diagnostic Test: NGS testing

INTERVENTIONS:
Diagnostic Test: NGS testing — NGS test will be performed

SUMMARY:
Title of the study A study to examine the value of broad agnostic NGS panel testing versus reimbursed organ-directed NGS: a Belgian Precision study of the BSMO in collaboration with the Cancer Centre Study Number BSMO 2020-1 Study Phase Exploratory Sponsor Belgian Society of medical Oncology (BSMO) Treatment None Background and Rationale Several drugs targeting mutated gene products in cancer cells are available to Belgian patients through reimbursement of the drugs and, soon, by reimbursed organ-specific genomic testing.

This context is unfavorable with regard to the following issues:

1. Many more additional drugs with sound scientific rationale and preclinical evidence are available through clinical trials. The relevant genes are generally not included in the reimbursed NGS and ad hoc identification of such patients is extremely difficult and thus severely hampering the accrual in such trials. This denies patients a potential access to innovative treatments from which they could benefit and hampers progress.
2. The same genes can be mutated in other cancer types, other than the reimbursed context, but are not detected due to the organ-specific approach in reimbursed NGS. Examination of these genes with an agnostic approach would give these other patients potential access to the drugs (via various routes, including clinical trials or medical need or otherwise)
3. The broader panels applied by some Belgian platforms (50-100 genes), sometimes in an agnostic approach, do not cover all potentially actionable genes or not all types of actionable variants in these genes.
4. Rearrangements which are highly actionable are not systematically covered in NGS testing, but rely on immunohistochemistry (if done at all) of fusion panels testing that requires additional funding.
5. The various Belgian NGS labs use accredited but heterogeneous methodology and it has been reported that the detection rate of some mutations varies from one site to another.

Therefore, from a patient and oncologist point of view there are current deficiencies that jeopardize optimal access of patients to current or novel genome-driven therapies. Defective identification of sensitive patients limits the implementation of clinical trials and their accrual rates and therefore the attractiveness of Belgium for such trials.

There are more comprehensive commercial platforms that cover a large set of actionable genes (up to hundreds of genes) and the various types of mutations in these genes: sequence mutations, rearrangements, resulting in fusion genes, and gene amplifications.

These commercial vendors have adequate comprehensive methodology but are too expensive (at their current public pricing) for general application. One of these is the platform of Foundation Medicine that builds on a large experience in variant annotation in the US and includes probably all current actionable targets including gene mutations, fusions, MSI, and TMB, all at once in one result. They also report actionability and established or clinical trial treatment options.

To oncologists this is very attractive compared to the fragmented, sequential and very limited current reimbursed conditions.

The investigators estimate that up to 20% of advanced cancer patients could get access to genotype-based treatment that are not covered by the organ-based reimbursement based access to NGS. This can be in the form of off-label application of reimbursed drugs, pharma-sponsored drug development trials that address a specific genotype or pharma sponsored or academic basket trials. Without broad agnostic testing the identification of eligible patients remains extremely difficult. A recent study [A study of genetic characteristics and suitability for targeted cancer treatment (TARGET)] showed that the rate of detection of actionable mutations increased from 28% with local testing to 66% with Foundation Medicine testing.

Objectives

1. To determine the added value of comprehensive and agnostic NGS versus "real-world" practice ("real-world" practice means local testing, no reimbursement for local testing and/or no accessible metastatic lesion) in providing patients with advanced/metastatic solid tumors access molecular guided therapy and/or immunotherapy based on genomic results.
2. To describe the landscape of genomic alterations detected by reimbursed NGS
3. To describe he landscape of genomic alterations detected by comprehensive panel testing
4. To assess the technical success of comprehensive panel testing
5. To describe the uptake of treatments recommended by the molecular tumor board guided by the genomic testing.

ELIGIBILITY:
Inclusion Criteria:

* 1- Adult patients (18 years and above)
* 2- Patients with metastatic solid tumors that are candidates for systemic therapy (early lines are preferred). Numbers will be capped for frequent tumor types (breast cancer: 150 patients, NSCLC: 150 patients, colorectal cancer: 150 patients). There will be a cohort of 200 patients with rare tumors or tumors with rare histology (Eur. J. Cancer 2011; 47: 2493-2511). Patients will be recruited as they appear in clinical practice.

  3- Patients will be enrolled following three clinical scenarios: a) patients eligible for local NGS testing (reimbursed or local practice); b) patients that are not eligible for reimbursed or local NGS testing; c) patients with no sufficient archival tissue meeting the pre-requirements will only undergo FMI liquid biopsy testing (exploratory cohort). That last cohort will be capped at 100 patients and will not have more than 50% of patients with the same tumor type.

  4- Patients enrolled in scenario a) and b) must have enough tissue from a metastatic (preferred) or primary lesion biopsy for local testing and FMI testing. The tissue should not be more than 3 years-old and fixed in 10% neutral buffered formalin. Availability of metastatic biopsies performed after a previous therapy line are mandatory for patients treated with therapies that are known to induce acquired mechanisms of resistance (EGFR TKIs in NSCLC, aromatase inhibitors in breast cancer, TKIs in Gastrointestinal stromal tumor (GIST)…). Bone biopsies that undergo decalcification are not allowed.

  5- Patient showing an Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 2.

  6- Patients can only be enrolled if they are also concomitantly registered in the Precision 1 study and the investigator agrees to subsequent registration of genotype-driven treatments given and the investigator assessed outcome on these treatments (RR and PFS).

  7- Patients able to provide written informed consent prior to enrollment into a potential subsequent clinical trial.

Exclusion Criteria:

* 1- Life expectancy of less than 12 weeks.
* 2- Inability to comply with protocol procedures.
* 3- Known presence of severe hematopoietic, renal, and/or hepatic dysfunction (according to the local PI).

  4- - No informed consent provided.
* 5- Patient is not enrolled and followed as provided in Precision 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2020-10-09 (Actual); Primary Completion 2022-09-15 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Number/prevalence of level 1, 2, 3 and 4 alterations as per OncoKB using comprehensive panel testing versus "real-word" practice in the three cohorts included. | through study completion, an average of 1 year
Number/prevalence of alterations by type using Foundation Medicine testing. Descriptive results will also be presented by tumor type. | through study completion, an average of 1 year
Percentage of patients with successful comprehensive panel testing | through study completion, an average of 1 year

SECONDARY OUTCOMES:
Prevalence of level 1, 2, 3 and 4 alterations as per OncoKB detected using liquid biopsies. | through study completion, an average of 1 year
Percentage of patients with a treatment recommandation based on a liquid biopsy | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (12):
- Belgium (12):
  - ZNA, Antwerp
  - GZA, Antwerp
  - AZ Klina, Brasschaat
  - Institute Jules Bordet, Brussels
  - AZ VUB, Brussels
  - Les Cliniques Universitaires St Luc, Brussels
  - Grand Hôpital de Charleroi, Charleroi
  - Universitaire Ziekenhuis Antwerpen, Edegem
  - UZ Gent, Ghent
  - Jessa Ziekenhuis, Hasselt
  - CHU Sart-Tilman, Liège
  - AZ Nikolaas, Sint-Niklaas

IPD SHARING:
Plan to Share IPD: Undecided